CLINICAL TRIAL: NCT00084123
Title: Healing Touch in Advanced Cervical Cancer Patients: Immune Effects and Mechanisms
Brief Title: Healing Touch and Relaxation Therapies in Cervical Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P20AT000756-01 (NIH); NCT00065091 (obsolete NCT alias)
Record Dates: First submitted 2004-06-07; First posted 2004-06-08 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Cervix Neoplasms
Keywords: Relaxation Techniques; Radiation; Drug Therapy; Healing Touch
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Relaxation Therapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healing Touch (Experimental): Healing Touch Therapy
  Interventions: Behavioral: Healing Touch Therapy
- Relaxation Therapy (Active Comparator): Relaxation Therapy
  Interventions: Behavioral: Relaxation Therapy
- Standard Care (Placebo Comparator): Standard Care
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Healing Touch Therapy
  Arms: Healing Touch
Behavioral: Relaxation Therapy
  Arms: Relaxation Therapy
Behavioral: Standard Care — Standard Care
  Arms: Standard Care

SUMMARY:
The purpose of this study is to evaluate the effects of healing touch and relaxation therapy on cervical cancer patients undergoing chemotherapy and radiation treatment.

DETAILED DESCRIPTION:
The side effects of chemotherapy and radiation treatment are often severe and can have devastating effects on the mental and physical well-being of cancer patients. This study will determine whether healing touch and relaxation therapy are effective in minimizing the side effects of chemotherapy and radiation treatment in cervical cancer patients.

Participants in this study will receive weekly chemotherapy and daily radiation treatments for 6 weeks. Participants will be randomly assigned to receive either standard care (SC), SC plus relaxation therapy, or SC plus healing touch therapy. The relaxation therapy consists of progressive muscle relaxation and guided imagery. The healing touch therapy involves an energy-based modality in which health care practitioners stimulate the energy fields surrounding the patient. A physician-completed assessment and measures of immune function will be used to assess the well-being and overall quality of life of participants.

ELIGIBILITY:
Inclusion Criteria:

* Stage Ib1-IVa cervical cancer
* Treatment with concurrent chemotherapy and radiation at the University of Iowa Hospitals and Clinics

Exclusion Criteria:

* Immunosuppressive disorders
* Use of immunosuppressive medications
* Transplant recipient
* Metastatic or recurrent cervical cancer
* History of any other type of cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
natural killer cell cytotoxicity | Baseline to week 6
T-cell counts | Baseline to week 6
side effects | Baseline to week 6

SECONDARY OUTCOMES:
distress | Baseline to week 6
WBC and RBC | Baseline to week 6
days of treatment delay | Baseline to week 6
salivary cortisol | Baseline to post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Susan K Lutgendorf, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospital and Clinics, Iowa City, Iowa, United States